CLINICAL TRIAL: NCT05797324
Title: Multicenter Study on the Role of Light Therapy in Modulating the Clinical Phenotype of Patients With Primary and Comorbid Chronic Insomnia Through Circadian Phase Modification.
Brief Title: Light Therapy in Modulating the Clinical Phenotype of Patients With Primary and Comorbid Chronic Insomnia.
Acronym: Luminoterapia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Ente Ospedaliero Cantonale, Ticino, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21A011
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Insomnia Chronic
Keywords: Light therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luminette (Experimental): Patients without ocular contraindications undergo a Luminotherapy protocol (intermittent blue-enriched light therapy with Luminette 10000 lux equivalent) with morning or evening timing, depending on the circadian phase.
  Interventions: Other: Luminette
- Sham (Sham Comparator): Control group (white light <100 lux equivalent).
  Interventions: Other: Sham

INTERVENTIONS:
Other: Luminette — Luminotherapy protocol (intermittent blue-enriched light therapy with Luminette 10000 lux equivalent) with morning or evening timing, depending on the circadian rhythm
  Arms: Luminette
Other: Sham — Sham protocol (white light <100 lux equivalent).
  Arms: Sham

SUMMARY:
Some evidence indicates that circadian rhythm may play a role in the pathophysiology of insomnia disorder. This single-blind randomized controlled multicentre prospective study aims to evaluate the possible therapeutic effect of light therapy in modulating the clinical phenotype of patients affected by chronic primary and comorbid insomnia, through the modification of the circadian phase.

DETAILED DESCRIPTION:
Some evidence indicates that circadian rhythm may play a role in the pathophysiology of insomnia disorder. This single-blind randomized controlled multicentre prospective study aims to evaluate the possible therapeutic effect of light therapy in modulating the clinical phenotype of patients affected by chronic primary and comorbid insomnia, through the modification of the circadian phase.

STUDY DESIGN AND METHODS

With regard to the study in question, it should be noted that:

* the study is a prospective multicentre randomized single-blind controlled trial
* the duration of the study is expected to be 3 years with a duration of enrollment of 2 and a half years and a minimum clinical follow-up of 3 months

The study will be divided into two evaluations, an initial evaluation (Time 0, T0) where the patients will be enrolled and all the measurements required before treatment with light therapy will be performed, and a final evaluation after 6 weeks of treatment with light therapy effective or sham (Time 1, T1), where the measurements performed at T0 will be repeated. Both assessments will be performed at the Sleep Medicine outpatient clinic.

TIME T0

* The diagnosis of primary chronic or comorbid insomnia will be made during the semi-structured sleep interview by a physician expert in sleep medicine, according to DSM V criteria, supported by clinical scales (Insomnia Severity Index, Pittsburgh Quality Index). The presence of mood/behavioral disorders or cognitive deficits will also be excluded (Beck, Stai, Mini Mental Scale Examination).
* A home polysomnography will be performed to rule out the presence of sleep apnea disorder or periodic limb movement syndrome during sleep
* Circadian parameters (chronotype, Mid sleep, circadian phase, phase angle) will be evaluated in basal conditions through clinical scales (Morning Eveningness Questionnaire, Light diet), measurement of salivary melatonin using evening 5-point wipes at home (DLMO, Elisa) and the actigraphic registration extended for 7 days.
* The associations between the circadian phase and the various phenotypes of primary or comorbid insomnia will be then evaluated, according to the duration and the severity of insomnia.
* Patients without ocular contraindications will then undergo a Luminotherapy protocol (intermittent blue-enriched light therapy with Luminette 10000 lux equivalent) with morning or evening timing, depending on the circadian phase, or sham treatment (control subgroup; white light <100 lux equivalent).
* Patients will be randomly assigned to one of two conditions (treatment and sham). The randomization list will be generated with a simple randomization method through the use of a "Random number generator" software available at www.regione.emilia-romagna.t/sin_info/generatore. The algorithm used in this site coincides with a Lehmer generator (multiplicative congruential generator). Allocation concealment is guaranteed by a central randomization in a distant and independent location with respect to the recruitment site.

TIME T1

> After 6 consecutive weeks of home light therapy, patients will be re-evaluated with the same somnometry battery used at study entry. Furthermore, the actigraphic monitoring and the dosage of salivary melatonin will be repeated, to evaluate the variations of the circadian phase and of the sleep-wake pattern after light therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary chronic insomnia
* Comorbid chronic insomnia
* Absence of pharmacological therapy of insomnia
* Absence of behavioural and cognitive treatment of insomnia
* Capacity to understand the study and adhere to the procedures
* Written informed consent

Exclusion Criteria:

* Secondary insomnia due to medical conditions or drug treatment
* Cerebral diseases
* Invalidating diseases
* Eye diseases that contraindicate the use of light therapy
* Psychiatric disorders
* Cognitive decline
* Working in night shifts during the last month before enrolment
* Impossibility to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Baseline and after 6 weeks of intervention
  Insomnia Severity Index (ISI, Pittsburgh Quality Index) - self-report questionnaire composed of 19 items assessing sleep quality

SECONDARY OUTCOMES:
Change in salivary melatonin | Baseline and after 6 weeks of intervention
  Salivary melatonin - evening 5-point wipes (DLMO, Elisa)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Oggebbio, Italy